CLINICAL TRIAL: NCT04585282
Title: A Randomized Controlled Study of Cognitive Behavioral Therapy for Insomnia With Anxiety and Depression
Brief Title: CBT for Insomnia With Anxiety and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chengmei Yuan
Record Dates: First submitted 2020-09-09; First posted 2020-10-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-07

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: In this study, patients were randomly assigned to study group and control group by random number table.
Who Masked: Investigator
Masking Description: The blind method of this study is evaluator blindness, that is, the evaluator does not know the grouping of subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The study group was treated with intensive cognitive behavioral therapy for insomnia.
  Interventions: Behavioral: Plus Cognitive behavioral therapy of insomnia（CBT-I plus）
- control group (Active Comparator): The control group was treated with traditional cognitive behavioral therapy for insomnia.
  Interventions: Behavioral: Cognitive behavioral therapy of insomnia（CBT-I）

INTERVENTIONS:
Behavioral: Plus Cognitive behavioral therapy of insomnia（CBT-I plus） — Cbt-i plus program is an enhanced version of cbt-i program, which increases the response to depression and anxiety symptoms.
  Arms: intervention group
Behavioral: Cognitive behavioral therapy of insomnia（CBT-I） — Cognitive behavioral therapy of insomnia is mainly aimed at correcting the bad behaviors and beliefs among the maintenance factors of insomnia, which is considered as the first-line treatment program of insomnia disorder. Cognitive behavioral therapy of insomnia mainly includes five important components: sleep restriction, secondary control, cognitive therapy, relaxation therapy and sleep hygiene.
  Arms: control group

SUMMARY:
Objective to explore whether cbt-i plus is more effective and feasible for patients with insomnia complicated with anxiety and depression than the traditional cognitive behavioral therapy for insomnia.

Hypothesis: cbt-i plus is superior to cbt-i in efficacy and feasibility.

DETAILED DESCRIPTION:
The purpose of this study was to explore the treatment of cognitive behavioral enhancement of insomnia (cbt-i plus), which was randomly divided into cbt-i plus intervention group (Study Group) and cbt-i intervention group (control group). The study group used the unified cognitive behavioral therapy manual for insomnia (cbt-i plus) for one-to-one individual treatment intervention, once a week, 45-50 minutes each time, a total of 8 times; the control group used the unified cognitive behavioral therapy manual for insomnia (cbt-i) for one-on-one treatment intervention, once a week, 45-50 minutes each time, a total of 8 times. The related indexes were evaluated at baseline, 2 weeks, 4 weeks and 8 weeks after enrollment, and were followed up at 12 weeks and 24 weeks after enrollment. Hypothesis: cbt-i plus is superior to cbt-i in efficacy and feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male and female
2. Meet the diagnostic criteria of DSM-5 for insomnia, the Pittsburgh Sleep Quality Index (PSQI) scale total score ≥10
3. May be accompanied by depression symptoms, but currently does not meet any depression disorders diagnostic criteria,14≤HAMD-17≤23
4. May be accompanied by anxiety symptoms, but currently does not meet any anxiety disorders diagnostic criteria ,14≤HAMA≤29
5. Have sufficient education and understanding to complete this study to be examined and evaluated
6. Voluntary participation in this clinical trial and signature of informed consent.

Exclusion Criteria:

1. DSM-5 other sleep problems, such as apnea syndrome, restless leg syndrome
2. Women who are pregnant, nursing or planning to become pregnant during the study
3. Insomnia caused by alcohol or substance abuse
4. Severe cognitive problems
5. Patients who were previously or currently diagnosed as bipolar and related disorders, obsessive-compulsive and related disorders, schizophrenia spectrum and other psychotic disorders, trauma and stress related disorders, separation disorders, eating disorders
6. Patients with history of epilepsy or other serious somatic diseases
7. Persons receiving MECT treatment for nearly one month
8. Excluding those who have received systemic psychotherapy for more than 3 months in a row
9. The researchers believe that it is not suitable to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of sleep efficiency | Change from Baseline Sleep efficiency at 8 weeks
  Sleep efficiency was measured by sleep diary
  Sleep efficiency was measured by sleep diary
Change of depressive symptoms | Change from Baseline Sleep efficiency at 8 weeks
  The measurement tool is Hamilton Depression Scale-17 items,the minimum score of the scale was 0 and the maximum score was 52. The higher the score was, the more serious the depression was.
Change of anxiety symptoms | Change from Baseline Sleep efficiency at 8 weeks
  The measurement tool is Hamilton Anxiety Scale,
  the minimum score of the scale was 0 and the maximum score was 56. The higher the score was, the more serious the anxiety was.

CONTACTS AND LOCATIONS:
Overall Officials: Chengmei Yuan, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No